CLINICAL TRIAL: NCT00739323
Title: Impaired Wound Healing in Diabetic Foot Ulceration
Acronym: EPC
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Aristidis Veves, Rongxiang Xu, MD Professor of Surgery in the Field of Regenerative Therapeutics, Beth Israel Deaconess Medical Center
Other Study IDs: 2006P000335; R01DK076937 (NIH); 1R01DK076937 (NIH)
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An observational study to gather information about people who may have certain abnormalities in skin microcirculation and muscle metabolism and to determine whether these abnormalities affect wound healing. The study also examines the association of a specific type of cell with the rate of wound healing.

DETAILED DESCRIPTION:
An observational study which entails: medical history; physical examination; blood tests; MRI; microcirculation tests (two noninvasive tests: 1) a procedure that measures the resting blood flow of the skin and 2) a technique that introduces acetylcholine and sodium nitroprusside in the skin and measures the ability of the skin's vessels to dilate and increase blood flow); and macrocirculation tests (noninvasive ultrasound of arm). This study also involves 2 Visits to the Beth Israel Deaconess Medical Center in Boston, MA. (Joslin-Beth Israel Deaconess Foot Center, Lowry Outpatient Laboratory, MRI Suite).

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Type I or Type II Diabetes Mellitus.
* Ulcer present for minimum 4 weeks
* Have adequate circulation to the foot
* Can return for follow-up visits
* Be able to read and sign the Informed Consent form before enrollment

Exclusion Criteria:

* Active Charcot's foot ulcer on the foot to be studied
* Presence of any serious disease that can affect wound healing including end stage renal failure requiring hemodialysis or renal transplantation, active malignant disease requiring treatment, hepatic, hematologic, neurologic, or immune disease
* Alcohol or drug abuse problems
* Treatment with oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents
* Presence of infectious disease that can preclude EPC measurements (including HIV, Hepatitis B and C)
* Pregnancy

Ages: 21 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects may be selected from the Beth Israel Deaconess Foot Clinic or from the Boston area and surrounding locations.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2006-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aristidis Veves, DSc, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States